CLINICAL TRIAL: NCT07062900
Title: Effects of Low Intensity Physical Activity on Functional Capacity Quality of Life and Psychological Well Being in Congestive Heart Failure Patients Among Different BMI
Brief Title: Low Intensity Physical Activity in Congestive Heart Failure Patients Among Different BMI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0360
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
Keywords: Congestive Heart Failure, low intensity Physical Activity, functional capacity, quality of life, psychological well-being, Body Mass Index.
MeSH Terms: conditions — Heart Failure; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Intensity Physical Activity Group (Experimental): Participants in this group underwent an 8-week structured low-intensity physical activity program. The program included gentle walking, use of a portable pedal exerciser, light resistance band exercises, and functional activities like seated leg press and hip circles. Sessions gradually increased in duration and frequency, starting from 2 sessions per week to 3 sessions per week, lasting 20-40 minutes each. The focus was on improving functional capacity, psychological well-being, and quality of life without causing cardiac stress.
  Interventions: Behavioral: Low-Intensity Physical Activity; Behavioral: usual care
- Usual Care Group (Active Comparator): Participants in this group received standard medical care only, with no additional structured physical activity or intervention. They continued their routine treatment and lifestyle without any specific exercise regimen. This group served as the comparison group to evaluate the effects of the physical activity intervention.
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: Low-Intensity Physical Activity — This includes a structured and progressive 8-week physical activity program involving:
  Gentle walking
  Portable pedal exerciser
  Low-intensity resistance exercises (e.g., resistance bands, seated leg press, hip circles)
  Supervised sessions with warm-up and cool-down components
  Arms: Low-Intensity Physical Activity Group
Behavioral: usual care — Standard Medical Management: Participants continued with their prescribed medications and routine clinical follow-ups for congestive heart failure as directed by their healthcare providers.

SUMMARY:
This study examined the effects of low-intensity physical activity on functional capacity, quality of life, and psychological well-being in congestive heart failure patients with varying BMI. Forty patients were divided into intervention and control groups. The intervention group followed an 8-week physical activity program, while the control group received usual care. Results showed significant improvement in walk distance, quality of life, and depression scores in the intervention group. The study concludes that low-intensity physical activity effectively improves health outcomes in heart failure patients across different BMI categories.

DETAILED DESCRIPTION:
This randomized controlled trial explored the effects of low-intensity physical activity on functional capacity, quality of life, and psychological well-being in patients with congestive heart failure across different BMI categories. A total of forty patients were selected and randomly assigned to either an intervention group or a control group. The intervention group participated in an eight-week structured low-intensity physical activity program, while the control group continued with usual care without additional physical activity. Various assessment tools were used to evaluate outcomes, including the 6-minute walk test to measure functional capacity, the Kansas City Cardiomyopathy Questionnaire to assess quality of life, and the Hospital Anxiety and Depression Scale to evaluate psychological well-being. The results demonstrated that although both groups showed some improvement, the intervention group experienced significantly greater gains in all measured outcomes. The 6-minute walk distance increased, KCCQ-12 scores improved notably, and depressive symptoms reduced significantly in the intervention group compared to the control. The study concluded that low-intensity physical activity is an effective and feasible intervention to enhance physical and mental health in congestive heart failure patients, irrespective of their BMI category.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized Congestive heart failure patients
* Age 45-70
* Diagnosed with CHF
* BMI all ranges
* Severely underweight: BMI<16 kg/m2
* Underweight: BMI≥ 16 kg/m2 and <18.5 kg/m2
* Normal weight BMI≥18.5 kg/mg2 and <25kg/m2
* Overweight: BMI ≥25kg/m2 and<30 kg/m2
* Obese: BMI≥30 kg/m2
* Willing to participate in physical activity program

Exclusion Criteria:

* Musculoskeletal or neurological disorders
* Severe COPD or other respiratory diseases
* Cognitive impairment
* Cardiac catheter related surgery, valvular surgery within past 6 month
* Recent Lung embolis
* Lung cancer
* Participants in other clinical trial or intervention study

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walk Test (6MWT) | 8 weeks
  Functional Capacity
Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 8 weeks
  Quality of Life
Hospital Anxiety and Depression Scale (HADS) | 8 weeks
  Psychological Well-Being

CONTACTS AND LOCATIONS:
Overall Officials: Arjumand Bano, Ms CPPT, Principal Investigator — Riphah International University
Locations (1):
- Arjumand, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No